CLINICAL TRIAL: NCT05713136
Title: The National Australian HCV Point-of-Care Testing Program: An Observational Cohort Study to Evaluate the Use of Finger-stick Point-of-care Hepatitis C Testing to Enhance Diagnosis and Treatment of HCV Infection - HCV Antibody Testing Minimal Dataset
Brief Title: The National Australian HCV Point-of-Care Testing Program - HCV Antibody Testing Minimal Dataset
Status: Recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Flinders University (Other)
Responsible Party: Sponsor
Other Study IDs: VHCRP2203
Record Dates: First submitted 2023-01-17; First posted 2023-02-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Hepatitis C
Keywords: Point-of-Care; Rapid Diagnostic Testing; HCV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People at risk of HCV acquisition: Clinic staff will offer HCV point-of-care testing to participants as they access services. Testing will be performed using point-of-care HCV RNA testing
  Interventions: Device: Diagnostic Test: Point-of-Care Testing

INTERVENTIONS:
Device: Diagnostic Test: Point-of-Care Testing — Participants will be offered finger-stick point-of-care testing for HCV

SUMMARY:
The goal of this observational study is to learn if offering a point-of-care screening test for exposure to the Hepatitis C virus, before providing a diagnostic test for Hepatitis C infection can increase testing, diagnosis and treatment in Adults. Participants will be recruited from settings that provide services to people with a risk factor for the acquisition of Hepatitis C viral infection. The main question it aims to answer is:

What proportion of the participants that have been diagnosed with HCV infection have started treatment when their records are reviewed 12 weeks after diagnosis?

Participants will have one in-person visit where they will provide informed consent and receive a finger-prick rapid result test for Hepatitis C infection. Participants with no previous Hepatitis C infection will have a screening test to see if they have an immune reaction to Hepatitis C. Participants who know they have been infected with Hepatitis C in the past, and all participants with a positive screening test result will then be given a Hepatitis C diagnostic test at this visit.

No treatment is provided as a part of this study, participants who are diagnosed with Hepatitis C infection will be referred to testing locations standard of care for any additional clinical assessments and treatment initiation. A review of the participant's records will be made 12 weeks after their Hepatitis C result and their treatment data are gathered.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* ≥ 18 years of age.

Exclusion Criteria:

* Is unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be included from settings that provide services to people with a risk factor for the acquisition of HCV infection, including drug treatment clinics, needle and syringe programs, prisons, mobile outreach services, community health services, mental health services, homelessness services, and other appropriate settings nationally. It is anticipated that approximately 40,000 participants will be screened for HCV infection using point-of-care HCV testing.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of HCV infected (HCV RNA quantifiable) participants who initiate HCV treatment at 12 weeks following finger-stick point-of-care HCV RNA testing. | 12 weeks from enrolment
  HCV treatment

SECONDARY OUTCOMES:
To evaluate the proportion of people who accept point-of-care testing among those offered testing. | Recruitment phase
  Accepting testing
To evaluate the prevalence of current HCV infection (HCV RNA quantifiable) among people tested. | Recruitment phase
  Prevalence
To evaluate the HCV antibody prevalence among people tested. | Recruitment phase
  Prevalence
To evaluate the time to treatment uptake among people receiving point-of-care HCV antibody testing with reflex HCV RNA testing in those who are HCV antibody detectable who received HCV treatment; | 52 weeks
  Time to treatment
To evaluate the proportion of HCV RNA positive participants who initiate HCV treatment at 12 months (52 weeks) following finger-stick point-of-care HCV RNA testing. | 52 weeks
  Initiation of treatment
To evaluate the proportion of participants who complete HCV direct-acting antiviral (DAA) treatment following point-of-care HCV antibody testing with reflex HCV RNA testing in those who are HCV antibody detectable who received HCV treatment; | 52 weeks
  Completion of treatment
To evaluate the proportion of participants who achieve an SVR following point-of-care HCV antibody testing with reflex HCV RNA testing in those who are HCV antibody detectable who received HCV treatment | 52 weeks
  SVR
To evaluate the proportion of participants who are HCV RNA negative at 12 months (52 weeks) following finger-stick point-of-care HCV RNA testing. | 52 weeks
  HCV negative
To evaluate the cost of point-of-care HCV antibody testing prior to reflex HCV RNA testing compared to direct point-of-care HCV RNA testing and standard of care. | 52 weeks
  Cost-effectiveness

CONTACTS AND LOCATIONS:
Locations (12):
- Australia (12):
  - ACT Justice Health, Canberra, Australian Capital Territory
  - Justice Health and Forensic Mental Health Network, Sydney, New South Wales
  - Queensland Injectors Health Network Ltd, Bowen Hills, Queensland
  - West Moreton Hospital and Health Service, Brisbane, Queensland
  - Lotus Glen Correctional Centre, Cairns, Queensland
  - Townsville Correctional Centre, Townsville, Queensland
  - Woodford Correctional Centre, Woodford, Queensland
  - South Australian Prison Health Service, Adelaide, South Australia
  - Hepatitis South Australia, Hackney, South Australia
  - Tasmanian Prison Service, Hobart, Tasmania
  - St Vincent's Hospital (Melbourne), Melbourne, Victoria
  - WA Department of Justice, Perth, Western Australia

DOCUMENTS (1):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT05713136/Prot_000.pdf